CLINICAL TRIAL: NCT01208870
Title: Translating Habituation Research to Interventions for Pediatric Obesity
Acronym: EAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Leonard Epstein, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1083316-1-52205; 5U01DK088380 (NIH)
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Pediatric Obesity; Habituation
MeSH Terms: conditions — Pediatric Obesity; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Variety Group (Experimental): Traditional family based weight control treatment program with components to reduce variety of high energy dense foods incorporated into the treatment. Families meet weekly for 12 weeks, then by-weekly for 1 month and 1 monthly session for a total of 15 behavioral intervention sessions.
  Interventions: Behavioral: Variety Group; Behavioral: Nutrition Education Control
- Nutrition Education Control (Experimental): Traditional family based weight control treatment program, without components from habituation theory incorporated into the treatment. Families meet weekly for 12 weeks, then by-weekly for 1 month and 1 monthly session for a total of 15 behavioral intervention sessions.
  Interventions: Behavioral: Nutrition Education Control

INTERVENTIONS:
Behavioral: Variety Group — The intervention will consist of our traditional family based weight control intervention with elements of reducing variety of high energy dense foods for the variety group.
  Arms: Variety Group
Behavioral: Nutrition Education Control — The intervention will consist of our traditional family based weight control intervention.

SUMMARY:
The purpose of this center grant is to translate basic behavioral science on habituation theory into clinical intervention using a vertical hierarchical approach from laboratory studies to field studies to the clinical intervention to improve weight loss outcomes in pediatric obesity treatment.

DETAILED DESCRIPTION:
Habituation is one factor that may be related to excess energy intake. Research has shown that the rate of habituation is inversely related to the amount of food consumed and slower habituation may be a factor that is relevant to obesity, as overweight youth and adults habituate slower and consume more energy than their peers. Habituation is a basic form of learning that is observed in many response systems. We believe that habituation is an important process that mediates food regulation during a meal and across meals. However, there has been no research in children that translates basic research on habituation to food into clinical interventions for pediatric obesity. In the first phase, we will implement a series of laboratory studies to assess the effects of stimulus specificity and variety and the simultaneous reduction of variety for high energy density foods on short (within meal) and long-term (across meal) habituation. The second phase is designed to implement a series of field studies that will extend basic research from the first phase as well as define the optimal interval for reducing variety to facilitate long-term habituation to high energy density foods in the natural environment. The third phase is designed to develop and pilot test a family-based behavioral intervention for children that incorporates findings from phase2 into a clinical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8-12 years of age
* At or above 85th BMI percentile
* Children must eat almost all meals with the exception of school lunch with the family.
* Overweight parent

Exclusion Criteria:

* Children who do not like the study foods, who are allergic to the study foods or who are on special diets and cannot consume the study foods.
* Families with children with a co-morbid psychiatric diagnosis or parents who are depressed, have schizophrenia, substance abuse or a history of eating disorders.
* The parent and child must not have any physical restrictions that would preclude them from making the requisite behavioral changes.
* Children must be able to read at a 3rd grade reading level and must be able to demonstrate the ability to keep dietary and activity records in a stimulated interview.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2009-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard H. Epstein, Ph.D., Principal Investigator — SUNY Buffalo
Locations (1):
- University at Buffalo, Department of Pediatrics, Division of Behavioral Medicine, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared under the specifics of this protocol. Outcome data will be published.

REFERENCES:
- [Derived] Epstein LH, Kilanowski C, Paluch RA, Raynor H, Daniel TO. Reducing variety enhances effectiveness of family-based treatment for pediatric obesity. Eat Behav. 2015 Apr;17:140-3. doi: 10.1016/j.eatbeh.2015.02.001. Epub 2015 Feb 13. PMID 25706950
- [Derived] Epstein LH, Fletcher KD, O'Neill J, Roemmich JN, Raynor H, Bouton ME. Food characteristics, long-term habituation and energy intake. Laboratory and field studies. Appetite. 2013 Jan;60(1):40-50. doi: 10.1016/j.appet.2012.08.030. Epub 2012 Oct 22. PMID 23085682
- [Derived] Epstein LH, Carr KA, Cavanaugh MD, Paluch RA, Bouton ME. Long-term habituation to food in obese and nonobese women. Am J Clin Nutr. 2011 Aug;94(2):371-6. doi: 10.3945/ajcn.110.009035. Epub 2011 May 18. PMID 21593492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in the Western New York area targeted obese and overweight families through pediatric offices and the local community during 2011-2013.
Pre-assignment Details: Interested eligible families are oriented, consented, screened, and offered to start the study. There were 94 participants (47 parents and 47 children) eligible to start and 4 participants (2 parents and 2 children) declined before starting the study.
Groups:
- Experimental Group: Traditional family based weight control program with components from habituation theory incorporated into the treatment.
  Habituation theory and Pediatric Obesity: The intervention will consist of our traditional family based weight control intervention with elements of habituation theory included for the experimental group. Experimental
- Nutrition Education Control: Traditional family based weight control program, without components of habituation theory incorporated.
  Habituation theory and Pediatric Obesity: The intervention will consist of our traditional family based weight control intervention with elements of habituation theory included for the experimental group.
Period: Overall Study
Arm/Group | Experimental Group | Nutrition Education Control
Started | 46 (The same group was run as Pilot 1 Spring 2012 and Pilot 2 Summer 2013) | 44 (The same group was run as Pilot 1 Spring 2012 and Pilot 2 Summer 2013.)
Pilot 1 | 20 | 22
Pilot 2 | 26 | 22
Completed | 44 | 36
Not Completed | 2 | 8
Not completed — Lost to Follow-up | 2 | 8

BASELINE CHARACTERISTICS:
Population: Families including an overweight child and parent.
Groups:
- Experimental Group: Traditional family based weight control program with components from habituation theory incorporated into the treatment.
  Habituation theory and Pediatric Obesity: The intervention will consist of our traditional family based weight control intervention with elements of habituation theory included for the experimental group.
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Nutrition Education Control | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Customized [Mean (Standard Deviation); unit: years]
  Parent Age n=23 Experimental, n=22 Control | 43.2 (6.6) | 43.0 (6.4) | 43.1 (6.4)
  Child Age n=23 Experimental n=22 Control | 10.6 (1.3) | 10.8 (1.4) | 10.7 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender (male/female)
  Participants
    Female | 35 | 33 | 68
    Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity (NIH/OMB) parent and child
  Participants
    Hispanic or Latino | 0 | 2 | 2
    Not Hispanic or Latino | 46 | 42 | 88
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 13 | 19
  White | 34 | 28 | 62
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 44 | 90
Child percent overweight (%) [Mean (Standard Deviation); unit: Percent overweight based on BMI charts] — Percent overweight or percent overBMI is calculated as %OverBMI= [(BMI - BMI at 50th percentile)/BMI at 50th percentile]*100. Population: The measure is for the children only
  Percent overweight based on BMI charts
    number analyzed (Participants) | 23 | 22 | 45
    (all) | 77.1 (40) | 71.8 (29.2) | 74.5 (33.6)
Child z-Body Mass Index [Mean (Standard Deviation); unit: [1] z-BMI see description] — The formula for calculating LMS z-BMI scores based on age and sex is LMS method z-BMI = ((BMI/M L) - 1))/(L*S), where BMI = an individual's BMI, M =the median BMI for age and gender, L = power in the Box-Cox transformation for age and gender, and S =standard deviation for age and gender (Kuczmarski et al., 2002). A reference is Z-score of 0 is equal to the mean. Negative z-scores indicate values lower than the average and positive numbers indicate values higher than the average." Population: Children only
  [1] z-BMI see description
    number analyzed (Participants) | 23 | 22 | 45
    (all) | 2.2 (0.4) | 2.2 (0.4) | 2.2 (0.4)
Parent Weight (lb.) [Mean (Standard Deviation); unit: pounds] — Population: Parents only
  pounds
    number analyzed (Participants) | 23 | 22 | 45
    (all) | 236.8 (48.7) | 232.5 (46.2) | 234.7 (47.0)
Parent Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: Parents only
  kg/m^2
    number analyzed (Participants) | 23 | 22 | 45
    (all) | 38.9 (8.2) | 37.2 (6.8) | 38.1 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Change of Child Body Composition
Description: Child percent overweight difference from baseline to 6 month. The formula used to derive weight loss percentage was weight lost at 6 months divided by starting weight, multiplied by 100.
Time Frame: Baseline to 6 months
Population: Children that completed the reported measures. Two children did not complete the body composition measures from the experimental groups and four children from the control group did not complete this measure.
Measure: Mean (Standard Error); unit: percentage of weight
Arm/Group | Experimental Group | Nutrition Education Control
Number analyzed (Participants) | 21 | 18
percentage of weight | -16.1 (13.5) | -13.3 (9.6)

2. Secondary Outcome: Change in Dietary Intake of Calories
Description: Energy intake was calculated for parents and children as the different from baseline to six months of calories consumed. The first pilot used the calories generated from the Food Frequency Questionnaire (FFQ) report however the second pilot used calories from 24 hour recalls based on the Center of Disease Control data base or food labels.
Time Frame: Baseline to 6 months
Population: Parents and children, three families did not complete the dietary measures.
Measure: Mean (Standard Deviation); unit: calories
Groups:
- Experimental Group: Traditional family based weight control treatment program with components from habituation theory incorporated into the treatment. Families meet weekly for 12 weeks, then by-weekly for 1 month and 1 monthly session for a total of 15 sessions.
  Habituation theory and Pediatric Obesity: The intervention will consist of our traditional family based weight control intervention with elements of habituation theory included for the experimental group.
- Nutrition Education Control: Traditional family based weight control treatment program, without components from habituation theory incorporated into the treatment. Families meet weekly for 12 weeks, then by-weekly for 1 month and 1 monthly session for a total of 15 sessions.
  Habituation theory and Pediatric Obesity: The intervention will consist of our traditional family based weight control intervention with elements of habituation theory included for the experimental group.
Arm/Group | Experimental Group | Nutrition Education Control
Number analyzed (Participants) | 40 | 34
calories
  Child change in calorie intake from FFQ | -716.5 (1046.6) | -730.6 (765.6)
  Parent change in calorie intake from FFQ | -916.0 (719.8) | -962.2 (764.6)
  Child change in calorie intake from 24 hr recall | -432.4 (396.1) | -230.3 (501.5)
  Parent change in calorie intake from 24 hr recall | -690.4 (488.3) | -501.9 (488.0)

3. Primary Outcome: Change Parent Body Composition
Description: Parent Body Mass Index (kg/m^2) difference from baseline to 6 months
Time Frame: Baseline to 6 months
Population: Parents
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Experimental Group | Nutrition Education Control
Number analyzed (Participants) | 23 | 18
kg/m^2 | -3.6 (2.5) | -3.1 (2.4)

4. Secondary Outcome: Change in Parent Delay Discounting
Description: Kirby, small, medium and large reinforcers. The Kirby monetary choice questionnaire will be used to measure implusivity in parents and children. Participants are presented with a set of 27 choices between smaller immediate rewards and larger delayed rewards. An estimate of the participant's discounting rate parameter can be made from the pattern of choices and participants who discount the value of the delayed rewards more steeply are said to be more impulsive as measured in K-values. (0.25 impulsive to 0.00016 not impulsive)
Time Frame: Baseline to 6 months
Population: Parents that completed this measure pre and post. Ten parents did not complete this post measure.
Measure: Mean (Standard Deviation); unit: k value
Arm/Group | Experimental Group | Nutrition Education Control
Number analyzed (Participants) | 18 | 17
k value
  Small reinforcer | 0.003 (0.023) | 0.032 (0.067)
  Medium reinforcer | -0.005 (0.033) | 0.020 (0.059)
  Large reinforcer | -0.003 (0.017) | 0.024 (0.069)

5. Secondary Outcome: Change in Child Delay Discounting
Description: Kirby, small, medium and large reinforcers. The Kirby monetary choice questionnaire will be used to measure impulsivity in parents and children. Participants are presented with a set of 27 choices between smaller immediate rewards and larger delayed rewards. An estimate of the participant's discounting rate parameter can be made from the pattern of choices and participants who discount the value of the delayed rewards more steeply are said to be more impulsive as measured in higher K-values (0.25 vs 0.00016).
Time Frame: Baseline to 6 months
Population: Children that completed this measure at pre and post time points. Eleven children did not complete the post measure.
Measure: Mean (Standard Deviation); unit: k value
Arm/Group | Experimental Group | Nutrition Education Control
Number analyzed (Participants) | 17 | 17
k value
  Small reinforcer | 0.017 (0.071) | 0.006 (0.060)
  Medium reinforcer | 0.030 (0.073) | 0.025 (0.095)
  Large reinforcer | 0.038 (0.082) | 0.021 (0.060)

6. Secondary Outcome: Changes in Variety Measures
Description: Variety of high energy density foods (RED) and low energy density foods (GREEN) were calculated from the Food Frequency Questionnaire (FFQ) for pilot 1 and 24 hour recalls (24-HR) for pilot 2. High energy dense food or Red foods are low in nutrient density. Most Red foods come from the Fats, Oils and Sweets groups and are to be used sparingly. Modified foods from the Fats, Oils, and Sweets group are still considered to be Red foods, even if their energy level is low. These foods contribute little nutrients to the diet and compete for consumption of healthier foods. Green foods are high in nutrient density and low in energy density. Most Green foods come from the fruit and vegetable groups. Serving sizes were based off the serving sizes used in United States Department of Agriculture (USDA) common serving sizes. Coding was based on the serving sizes of the specified food items and used to calculate the changes from baseline to six months.
Time Frame: Baseline to 6 months
Population: Parents and children were measured, three families did not complete the dietary measures.
Measure: Mean (Standard Deviation); unit: food items
Arm/Group | Experimental Group | Nutrition Education Control
Number analyzed (Participants) | 40 | 34
food items
  Child Fats, Oils, Sweets variety from FFQ | -12.5 (16.1) | -16.7 (18.0)
  Child Fruit variety from FFQ | -6.3 (34.7) | -11.3 (19.1)
  Child Vegetable variety from FFQ | -0.0 (21.4) | -8.0 (16.2)
  Parent Fat, Oil, Sweets variety from FFQ | -24.3 (17.3) | -22.2 (17.6)
  Parent Fruit variety from FFQ | 16.7 (27.1) | 20.3 (27.2)
  Parent Vegetable variety from FFQ | 13.5 (19.2) | 16.5 (18.5)
  Child Fats, Oils, Sweets variety from 24-HR | -9.7 (5.9) | -3.7 (5.9)
  Child Fruit variety from 24-HR | 0.5 (1.6) | 0.4 (0.8)
  Child Vegetable variety from 24-HR | 0.4 (0.8) | -0.3 (0.5)
  Parent Fats, Oils, Sweets variety from 24-HR | -11.2 (4.4) | -1.2 (9.8)
  Parent Fruit variety from 24-HR | 1.0 (1.6) | 0.5 (1.2)
  Parent Vegetable variety from 24-HR | -0.1 (1.6) | 0.3 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected at baseline, each treatment session of 12 weekly, 4 by-weekly, 1 monthly and 6 months.
Description: 0 references the number of adverse events
Arm/Group | Experimental Group | Nutrition Education Control
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44
Other Adverse Events (participants affected / at risk) | 0/46 | 0/44

LIMITATIONS AND CAVEATS:
Two different measures were used to assess variety and calorie intake.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No